CLINICAL TRIAL: NCT00242229
Title: A 6 Month, Open-Label Evaluation of the Long-Term Safety of DVS-233 SR in Elderly Outpatients With Major Depressive Disorder (MDD)
Brief Title: Study Evaluating DVS-233 SR in Elderly Outpatients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 3151A1-307
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
To evaluate the overall safety and tolerability profile of two dose levels of DVS-233 SR during 6 months of open-label treatment in elderly outpatients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients men and women aged 65 years or older.
* Mini Mental State Examination score of 24 or above.
* Subjects must have a primary diagnosis of MDD based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), single or recurrent episode, without psychotic features, on study day 1, if depressive symptoms for at least 30 days prior to screening visit and minimum screening and study day -1 (baseline) scores of 16 on the Hamilton Psychiatric Rating Scale for Depression (HAM-D17).

Exclusion Criteria:

* Significant risk of suicide based on clinical judgment, including common suicidal thoughts, and suicide being considered as a possible solution, even without specific plans or intention.
* Current (within 12 months of baseline) psychoactive substance abuse or dependence (including alcohol), manic episode, posttraumatic stress disorder, obsessive-compulsive disorder, or a lifetime diagnosis of bipolar or psychotic disorder as assessed by the modified Mini International Neuropsychiatric Interview (MINI). Current (within 12 months of baseline) generalized anxiety disorder, panic disorder, or social anxiety disorder as assessed by the modified MINI and considered by the investigator to be primary, causing a higher degree of distress or impairment than MDD. Presence (within 12 months of baseline) of a clinically important personality disorder (such as antisocial, schizotypal, histrionic, borderline, narcissistic). Presence of dementia.
* Depression associated with the presence of an organic mental disorder due to a general medical condition or a neurologic disorder.

Other exclusion applies.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term safety and tolerability of DVS SR in elderly outpatients with MDD.

SECONDARY OUTCOMES:
To evaluate the long-term response of subjects receiving DVS SR for the clinical global evaluation, functionality, general well-being, pain and absence of depressive symptoms (Hamilton Psychiatric Rating Scale for Depression 17-item score < or = 7).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer